CLINICAL TRIAL: NCT05930054
Title: Dentoskeletal Changes In The Transverse Dimension Using Tooth Bone-Borne Vs. Bone-Borne Expansion Appliances: A Prospective, Randomized, Double-Blind Clinical Study With Cone-Beam Computed Tomography
Brief Title: Dentoskeletal Changes In The Transverse Dimension Using Tooth Bone-Borne Vs. Bone-Borne Expansion Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ahmet Yağcı, PROFESSOR, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDH-2020-10444
Record Dates: First submitted 2023-06-12; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Transverse Maxillary Deficiency
Keywords: Maxillary expansion; CBCT; tooth-bone-borne; bone-borne

STUDY DESIGN:
Intervention Model Description: Eighteen patients were divided into 2 groups: TBB group (n = 9, 16.11 ± 0.59 years of age) and BB group (n = 9, 15.33 ± 1.22 years of age). CBCT scans were obtained before treatment and after 3 months of expansion. Transverse skeletal and dental expansion, alveolar and tooth inclination, and buccal alveolar bone thickness were evaluated in maxillary first premolars and molars. Paired t tests and independent-sample t tests were used to compare the expansion appliances.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tooth-bone-borne (TBB) group (Other): The TBB appliance was composed of a central expansion jackscrew (Dentarum), 4 tubes, 2 bands on the upper first molars to facilitate placement of the appliance, and 1.5-mm diameter stainless steel arms extending to the premolar teeth. Soldered stainless steel tubes (internal diameter: 2.0 mm; external diameter: 3.0 mm; length: 2.0 mm) served as guides for miniscrew placement. The size of the screws (PSM) was chosen as 1.8 mm in diameter and 11 mm in length, considering the 2 mm height of the tubes, 1 to 2 mm gap between the appliance and the palate surface, 1 to 2 mm gingiva thickness, and 5 to 6 mm length required for the bicortical placement of the screw in the bone.
  Interventions: Device: skeletal anchorage and rapid palatal expansion
- bone-borne (BB) group (Other): The BB appliance was composed of a central expansion jackscrew, 4 tubes as described in TBB group, and less acrylic used around it to adjust its position. In order to carry it to the mouth after preparation on the cast model, essix was used, which also included the patient's teeth
  Interventions: Device: skeletal anchorage and rapid palatal expansion

INTERVENTIONS:
Device: skeletal anchorage and rapid palatal expansion — Eighteen patients were randomly divided into 2 groups through a free randomization program (Random Allocation Software 2.0). Baseline demographic characteristics were matched in both groups. All appliances were fabricated by the same technician in the orthodontic lab. All individuals were treated by a single practitioner.

SUMMARY:
This study aimed to investigate the skeletal, dentoalveolar, and periodontal changes of tooth-bone-borne (TBB) and bone-borne (BB) appliances with identical miniscrew placement using cone-beam computed tomography (CBCT) in the post-pubertal growth spurt stage.

DETAILED DESCRIPTION:
Eighteen patients were divided into 2 groups: TBB group (n = 9, 16.11 ± 0.59 years of age) and BB group (n = 9, 15.33 ± 1.22 years of age). CBCT scans were obtained before treatment and after 3 months of expansion. Transverse skeletal and dental expansion, alveolar and tooth inclination, and buccal alveolar bone thickness were evaluated in maxillary first premolars and molars. Paired t tests and independent-sample t tests were used to compare the expansion appliances.

ELIGIBILITY:
Inclusion Criteria:

* With a unilateral or bilateral morphological lateral crossbite
* Whose first molars and premolars had completely erupted at pretreatment
* With maxillary constriction of more than 4 mm and less than 10 mm
* Who were going through the post-pubertal growth spurt stage based on hand-wrist radiographs

Exclusion Criteria:

* craniofacial anomalies
* compliance problems
* systemic or genetic disease
* previous orthodontic treatment history

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Nasal Changes | up to 1 year
  Nasal Width:Distance between right and left inner lateral limits of nasal cavity, parallel to the base of the nasal cavity, Nasal Floor Width :Width at widest portion of floor of the nose

SECONDARY OUTCOMES:
Maxillary Skeletal Changes | up to 1 year
  Maxillary width:Maxillary width tangent to nasal base at tooth level ,palatinal maxillary width:The distance between the inner cortical points of the palatinal bone
Dentoalveolar Changes | up to 1 year
  The palatal alveolar angle (PAA) is the angle between the lines created by drawing tangents to the right and left palatal alveolar plates

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet YAGCI, PROFESSOR, Study Director — Erciyes University faculty of dentistry
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University Faculty of Dentistry ,Department of Orthodontics, Kayseri, Kayseri̇
  - Erciyes University Faculty of Dentistry, Department of Orthodontics, Kayseri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lagravere MO, Major PW, Flores-Mir C. Skeletal and dental changes with fixed slow maxillary expansion treatment: a systematic review. J Am Dent Assoc. 2005 Feb;136(2):194-9. doi: 10.14219/jada.archive.2005.0141. PMID 15782523
- [Background] Carlson C, Sung J, McComb RW, Machado AW, Moon W. Microimplant-assisted rapid palatal expansion appliance to orthopedically correct transverse maxillary deficiency in an adult. Am J Orthod Dentofacial Orthop. 2016 May;149(5):716-28. doi: 10.1016/j.ajodo.2015.04.043. PMID 27131254
- [Background] Lee KJ, Park YC, Park JY, Hwang WS. Miniscrew-assisted nonsurgical palatal expansion before orthognathic surgery for a patient with severe mandibular prognathism. Am J Orthod Dentofacial Orthop. 2010 Jun;137(6):830-9. doi: 10.1016/j.ajodo.2007.10.065. PMID 20685540